CLINICAL TRIAL: NCT02249520
Title: Calibration of MR and PET-MR Imaging Protocols at the Cedars-Sinai Medical Center (CSMC) Biomedical Imaging Research Institute (BIRI) Research Imaging Core
Brief Title: Calibration of MR and PET-MR Imaging Protocols at RIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Daniel S. Berman, Principal Investigator/Chief Cardiac Imaging/Nuclear Cardiology, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35521
Record Dates: First submitted 2014-09-09; First posted 2014-09-25 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Coronary Artery Disease
Keywords: Magnetic Resonance Imaging; MRI; Positron Emission Tomography; PET; PET-MR; mMR
MeSH Terms: conditions — Neoplasms; Coronary Artery Disease | interventions — Molecular Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PET-MR imaging on Biograph mMR scanner (Other): Research PET-MR imaging on Biograph mMR scanner will be conducted immediately following administration of FDG for clinically approved scan. No additional radioisotope will be administered for the research scan.
  Interventions: Other: PET-MR imaging on Biograph mMR scanner
- MR-only imaging on Biograph mMR scanner (Other): Participants will undergo research MR-only imaging on Biograph mMR scanner.
  Interventions: Other: MR-only imaging on Biograph mMR scanner
- MR imaging on the Siemens Vida 3T MR scanner (Other): Participants will undergo research MR imaging on the Siemens MR scanner
  Interventions: Other: MR imaging on the Siemens Vida 3T MR scanner

INTERVENTIONS:
Other: PET-MR imaging on Biograph mMR scanner — Participants will undergo PET-MR imaging on the Biograph mMR scanner to evaluate the technical aspects of the total acquisition protocol directly post clinical administration of FDG, thus removing the requirement for additional radioisotope.
  Other Names: Siemens Biograph mMR; molecular imaging; PET-MR; mMR
  Arms: PET-MR imaging on Biograph mMR scanner
Other: MR-only imaging on Biograph mMR scanner — Participants will undergo MR-only imaging to test the technical aspects of the MR-only protocol on the Biograph mMR scanner. No drug administered.
  Other Names: Siemens Biograph mMR; PET-MR
  Arms: MR-only imaging on Biograph mMR scanner
Other: MR imaging on the Siemens Vida 3T MR scanner — Participants will undergo MR imaging to test the technical aspects of the MR protocol on the Vida MR scanner
  Other Names: MRI
  Arms: MR imaging on the Siemens Vida 3T MR scanner

SUMMARY:
This is a protocol to facilitate on-site calibration of the technical aspects of the Siemens Biograph mMR (molecular MR) Positron Emission Tomography-Magnetic Resonance (PET-MR) scanner and the 3T Siemens Vida MR scanner at the Cedars-Sinai Medical Center (CSMC) Biomedical Imaging Research Institute (BIRI) Research Imaging Core after scanner installation. The mMR is a FDA-approved standard clinical device (non-experimental) and will be used in accordance with clearance and approval from the FDA. The Vida is a state-of-the-art FDA approved scanner and will be clinically licensed within a short time.

DETAILED DESCRIPTION:
PET-MR Protocol on the Biograph mMR: This protocol requires the use of a radioisotope. To avoid administering radioisotope solely for the purposes of this calibration, we will recruit 20 patients from the clinical population at the S. Mark Taper Foundation Imaging Center at CSMC who are already receiving an isotope dose for their standard-of-care examination and are willing to be scanned at the Research Imaging Core on the same day right after their clinical exam. Subjects who are having a PET-MR after receiving FDG will have the same body part scanned as they did for clinical testing.

MR-only Protocol on the Biograph mMR:To set up MR-only protocols, we will enroll 20 volunteers for MR-only on the mMR scanner. This is a standard MR scan with no isotope involved. Those volunteers who are participating in the MR-only scan will have major body parts and organs scanned as needed for calibration.

MR imaging on the Siemens Vida 3T scanner: applications training is taking place and we will build clinical protocols in the future

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* For MR-PET calibration: Outpatient undergoing standard-of-care 18FDG-PET at S. Mark Taper Foundation Imaging Center at CSMC
* For MR-only calibration: Volunteers who are responding to approved advertising to volunteer at the BIRI Research Imaging Core for research MR

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Any contraindications to MR imaging.
* Any contraindication to MRI, including metallic implants (valve replacement, pacemaker, implantable cardiac defibrillator, metallic spine material), intracranial clips, metallic fragments in eyes, and claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
composite of measures of organ uptake, maximum target-to-background ratio and maximum standard uptake value as standard with FDG PET for maximum image quality for all standard protocols. | one day
  The mMR is a FDA-approved standard clinical device (non-experimental) and will be used in accordance with clearance and approval from the FDA. Results obtained from these tests will not be analyzed towards the end point of any study and will solely be used to finalize and calibrate the technical performance of the new scanner. All scans will be visually assessed for technique calibration.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Berman, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States